CLINICAL TRIAL: NCT01276028
Title: Acupuncture for Vasomotor Symptoms
Brief Title: Acupuncture in Menopause
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00014892
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Vasomotor Symptoms
Keywords: Acupuncture; Hot Flashes; Menopause; Vasomotor Symptoms
MeSH Terms: conditions — Hot Flashes | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): This group will start acupuncture treatments within 3 weeks of consent and continue to receive up to 20 treatments over a six month period. The number of treatments will be jointly determined by the participant and the acupuncturist.
  Interventions: Procedure: Acupuncture
- Waitlist (Other): This group of participants will be asked to wait 6 months and will then be allowed to receive acupuncture.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — For the Acupuncture group: Women will be eligible to receive from 1 to 20 treatments over a six month period. These women will receive an initial evaluation by a acupuncturist and will be given a Traditional Chinese Medicine (TCM) diagnosis as well as a recommended treatment schedule which they can then negotiate.
  Women in the waitlist group will not receive any acupuncture for 6 months. At the end of the 6 month period the participants will be allowed to begin the acupuncture treatments.

SUMMARY:
The primary purpose of this study is to determine the effectiveness of acupuncture for treating vasomotor and other symptoms associated with menopause as acupuncture is generally practiced in the "real world" setting and to obtain a comprehensive assessment of use patterns and symptom relief over time. This study will allow us to determine treatment patterns recommended by practicing acupuncturists, adherence to these treatments, and the effectiveness of different treatment patterns for reducing hot flashes. Results of this study will provide meaningful information to women in terms of number and frequency of acupuncture treatments likely to be needed to reduce hot flashes.

ELIGIBILITY:
Inclusion Criteria:

* Women experiencing on average 4 Hot Flashes a day
* Women aged 45-60
* Peri or Post menopausal Women (No periods for at least 3 months)

Exclusion Criteria:

* Women who have initiated CAM or non-CAM treatments for hot flashes in the last 4 weeks
* Women who have changed their dose of a CAM or non-CAM treatments for hot flashes in the last 4 weeks
* Women who have initiated antidepressants in the last 3 months
* Women who have changed their dose of an antidepressant in the last 3 months
* Women who have had acupuncture in the last 4 weeks
* Women who have received acupuncture from one of the study acupuncturists in the last 6 months will be excluded from the study
* Women who describe their health as fair or poor are excluded from the study
* Women who have a diagnosis of Hemophilia
* Relatives and Co-Workers of the treating acupuncturists

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Subjective Hot Flashes | Up to 14 months
  Hot Flashes will be monitored via daily diary. This diary will be filled out daily for the first six months (post randomization) of the study and then 1 week per month for the remaining 6 months of the study.

SECONDARY OUTCOMES:
Objective Hot Flashes | 3 days
  Objective hot flashes measured by skin conductance
Other Symptoms | Up to 14 months
Quality of Life | Up to 58 weeks
  Measures your quality of life over the last week

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Avis, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Chapel Hill Doctors, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Avis NE, Coeytaux RR, Isom S, Prevette K, Morgan T. Acupuncture in Menopause (AIM) study: a pragmatic, randomized controlled trial. Menopause. 2016 Jun;23(6):626-37. doi: 10.1097/GME.0000000000000597. PMID 27023860